CLINICAL TRIAL: NCT02983032
Title: Brief Behavioural Treatment for Insomnia (BBTI) in Family Carers of People With Dementia: a Feasibility Study
Brief Title: Brief Behavioural Treatment for Insomnia in Dementia Carers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16/WS/0252
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Dementia
Keywords: Caregivers; Insomnia
MeSH Terms: conditions — Dementia; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brief behavioural treatment for insomnia (BBTI) (Experimental): A behavioural therapy for improving symptoms of insomnia in older adults focussing on sleep-related behaviour such as napping and when a person gets up and goes to bed.
  Interventions: Behavioral: BBTI

INTERVENTIONS:
Behavioral: BBTI — 3 group sessions over 4 weeks

SUMMARY:
Background: between 50-74% of dementia carers report some sleep disturbance. However, relatively few studies have looked at psychological treatment for insomnia in this group. Dementia carers may be particularly at risk for suffering negative consequences from the impact of sleep loss on top of the stress of their carer role. Researchers have found that Brief Behavioural Treatment for Insomnia (BBTI) can be effective for improving symptoms of insomnia in older adults. BBTI focusses on sleep-related behaviour such as napping and when a person gets up and goes to bed.

Aims: this study aims to explore whether delivering group-based, Brief Behavioural Treatment for Insomnia (BBTI) to family carers of people with dementia is feasible, given that, to date, this has not yet been explored.

Who is eligible?: carers with insomnia who care for a family member with dementia and live with them at home are eligible for inclusion in this study.

What is involved for participants?: taking part will involve an initial telephone discussion with a researcher to check suitability. Participants will then meet the researcher for assessment. Assessment includes a sleep interview and completing some questionnaires. Participants will then be required to attend 3 group sessions of BBTI across the space of 4 weeks. After attending the BBTI group, participants will be asked to fill in some of the same questionnaires that they filled in during assessment and again 4 weeks later. Participants will also be invited to take part in a focus group to give feedback about the treatment and their overall experience of being in the study.

DETAILED DESCRIPTION:
This study will explore the feasibility of delivering adapted BBTI in a group setting to family carers of people with dementia. The study will be a feasibility study given that delivering BBTI to groups of dementia carers hasn't been done before. It is therefore necessary to explore, in essence, whether it is 'do-able'. In-line with this, the current study will be considering the following:

* How many eligible participants consent to participate in the study?
* How many carers stay in the study until the end?
* Do carers find BBTI an acceptable treatment, are they able to comply with treatment instructions, and what modifications might be required?
* Are any improvements in sleep observed?
* Are any improvements in anxiety, depression and carer burden observed? It is hypothesised that carers' sleep will improve over the course of the study. Specifically, it is hypothesised that there will be a reduction in scores on the Pittsburgh Sleep Quality Index (PSQI), an increase in scores on the Sleep Condition Indicator (SCI), and an improvement in sleep diary parameters (increased sleep efficiency, a reduction in sleep latency and a reduction in wake time after sleep onset) following participation in BBTI. Sleep efficiency is calculated by dividing time spent in bed divided by time actually asleep; sleep latency is the time it takes you to fall asleep and reduction in wake time after sleep onset is the total time you are awake during the night after you first fall asleep. Based on a calculation, the sample size required is estimated to be 11. Given that some participants may withdraw from the study the study will aim to recruit 15 participants.

Procedure Individuals who are caring for a family member with dementia will be given a Participant Invitation Letter by healthcare workers and advertisements will be place in relevant clinics. Those interested in finding out more will make contact with the research team, who will screen potential participants. Those meeting the criteria will be sent a Participant Information Sheet and invited to attend a baseline assessment appointment. At the initial assessment appointment, the researcher will answer any questions the person has about the study, the Participant Information Sheet, or the Consent Form. They will then be asked to fill in the Consent Form before starting the assessment. If they do not consent the assessment will not be initiated. If they do consent, then the researcher will proceed to completing the baseline assessment. This will include the semi-structured sleep interview and questions regarding physical and mental health. The following measures will also be administered: Alcohol Use Disorders Identification Test (AUDIT), Drug Use Disorders Identification Test (DUDIT), Pittsburgh Sleep Quality Index (PSQI), Sleep Condition Indicator (SCI), Hospital Anxiety and Depression Scale (HADS) and the Zarit Burden Interview (ZBI).

Participants will also be shown how to complete a sleep diary at this appointment and will be asked to complete this for the two weeks prior to the first session of BBTI. The baseline assessment appointment is expected to last between 45-60 minutes.

The intervention will be delivered across 3 group sessions and 1 telephone consultation over a period of 4 weeks, as follows:

Week 1 - 90 minute group session (allowing time to cover all the educational material and to give individual sleep instructions as well as a break and initial group introductions) Week 2 - Group session (max 45 mins) Week 3 - Phone call (approx. 15 minutes) Week 4 - Final group session (max 45 mins) Week 5 - Appointments for post-treatment assessment

There will be two group facilitators and groups will have a maximum of 5 participants. Participants will be asked to keep sleep diaries throughout the intervention period. At the beginning of each session, participants will also be asked to complete the Stanford Sleepiness Scale in order to monitor daytime sleepiness.

The following measures will be administered post-treatment and at 4 week follow-up: Pittsburgh Sleep Quality Index (PSQI), Sleep Condition Indicator (SCI), Hospital Anxiety and Depression Scale (HADS) and the Zarit Burden Interview (ZBI).

ELIGIBILITY:
Inclusion Criteria:

* Carer of person with dementia
* Live with person being cared for
* Meet Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria for insomnia disorder with the exception that carers not meeting the frequency criterion of 3 times per week or duration criterion of 3 months will still be included if frequency is at least twice per week and duration 2 months.
* competent in English language and have good basic literacy skills.

Exclusion Criteria:

* unstable, moderate to severe mental health issues (particularly Major Depressive Disorder and Bipolar Disorder)
* already receiving a psychological intervention
* untreated sleep disorders eg obstructive sleep apnoea, restless legs syndrome and periodic limb movement disorders.
* current serious medical condition, such as cancer or recent remission from cancer
* learning disability or a neurological condition (e.g. Multiple Sclerosis, Parkinson's disease, epilepsy)
* being investigated for or existing diagnosis of degenerative condition
* sleep problem primarily due to having to be awake during the night/early morning to respond to the needs of the person they care for

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Sleep quality | Baseline and four weeks post-intervention
  Change in Pittsburgh Sleep Quality Index (PSQI) score

SECONDARY OUTCOMES:
Sleep condition | Baseline and four weeks post-intervention
  Change in score from Sleep Condition Indicator (SCI)
Anxiety | Baseline and four weeks post-intervention
  Change in score from Hospital Anxiety and Depression Scale (HADS)
Burden | Baseline and four weeks post-intervention
  Change in score from the Zarit Burden Interview (ZBI)
Sleep efficiency | Baseline and four weeks post-intervention
  Change in sleep efficiency (calculated by dividing time spent in bed by time actually asleep)
Sleep latency | Baseline and four weeks post-intervention
  Change in sleep latency (the time taken to fall asleep)
Wake time after sleep onset | Baseline and four weeks post-intervention
  Change in total time you are awake during the night after you first fall asleep

CONTACTS AND LOCATIONS:
Overall Officials: Maria Gardani, PhD, Principal Investigator — University of Glasgow
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No